CLINICAL TRIAL: NCT03149809
Title: Behavioral or Solifenacin Therapy for Urinary Symptoms in Parkinson Disease
Acronym: BOSS PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N2293-I
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Overactive Bladder; Parkinson Disease
Keywords: Urinary incontinence; Parkinson disease; Overactive urinary bladder; Nocturia
MeSH Terms: conditions — Urinary Bladder, Overactive; Parkinson Disease; Urinary Incontinence; Nocturia | interventions — Solifenacin Succinate

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Non-Inferiority Trial
Who Masked: Outcomes Assessor
Masking Description: Blinded assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral therapy (Active Comparator): Pelvic floor muscle exercise-based behavioral therapy
  Interventions: Behavioral: Pelvic floor muscle exercise-based behavioral therapy
- Drug Therapy (Active Comparator): Daily solifenacin drug therapy
  Interventions: Drug: solifenacin

INTERVENTIONS:
Drug: solifenacin — Antimuscarinic bladder relaxant, antagonizes bladder muscarinic receptors
  Other Names: Vesicare
  Arms: Drug Therapy
Behavioral: Pelvic floor muscle exercise-based behavioral therapy — Multicomponent intervention including fluid management, constipation management and behavioral techniques incorporating pelvic floor muscle-exercise based urge suppression and self-monitoring to reduce overactive bladder symptoms
  Arms: Behavioral therapy

SUMMARY:
The impact of urinary symptoms in Parkinson disease (PD) extends beyond worsened well-being. Urinary symptoms common in PD, especially incontinence and nocturia, are major risk factors for falls likely due to the combination of urinary urgency and impaired mobility (and falls are a leading cause of mortality in PD), for spouse/caregiver stress due to decreased mutuality in the relationship, and for institutionalization, largely due to increased disability. Additionally, most medications currently recommended for urinary symptoms in PD are anticholinergic and have the potential to worsen the progressive cognitive and autonomic burdens of the disease. Veterans with PD are also more likely to rely solely on VA for their health care than Veterans without PD. Thus, optimizing the care of urinary symptoms for Veterans with PD becomes imperative, particularly for VA. Using a non-inferiority design, this proposal seeks to demonstrate the comparative effectiveness of pelvic floor muscle exercise-based behavioral therapy versus drug therapy to treat urinary symptoms in PD.

DETAILED DESCRIPTION:
The number of persons with Parkinson Disease (PD) in the United States is expected to double by 2030 as the population ages. Importantly, this increase in the prevalence of PD will have greater impact within the Department of Veterans Affairs (VA) because the Veteran population is older than the general population and Veterans with PD are more likely than those without PD to rely solely on VA for their health care. While PD is often characterized by the motor symptoms of the disease (tremor, bradykinesia, rigidity), non-motor symptoms such as urinary symptoms correlate more closely with impaired well-being as the disease progresses. However, the impact of urinary symptoms in PD extends beyond worsened well-being. The urinary symptoms of overactive bladder (OAB), including urgency, frequency, and nocturia, with or without urinary incontinence, are the most common urinary symptoms of PD. OAB symptoms are associated with falls (a cause of increased mortality in PD), with spouse/caregiver stress, and, ultimately with institutionalization, thus it is critical that we optimize the care of urinary symptoms for Veterans with PD.

Several studies suggest abnormal central nervous system processing of sensory input from bladder afferent nerves contributes to OAB symptoms in PD, possibly because of delayed recognition of bladder fullness. This mirrors findings in non-PD populations with OAB. In the non-PD OAB population, pelvic floor muscle contractions diminish bladder muscle contraction and recent evidence demonstrates that behavioral training with pelvic floor muscle exercises improves the cortical integration of bladder afferent signals. Pelvic floor muscle exercise-based behavioral therapy for OAB symptoms requires individuals to learn a motor skill and implement an adaptive behavioral strategy to delay the need to void. Because of its effectiveness compared to drug therapy, pelvic floor muscle exercise-based behavioral therapy is recommended first-line in men and women with OAB who do not have PD. However, the most recent clinical guidelines for the treatment of urinary symptoms in PD recommend treatment with anticholinergic drugs. While some anticholinergic drugs are effective in reducing symptoms of OAB, it is important to note that there is a glaring lack of an empirical evidence base to promote these drugs in the setting of PD given that they add to the anticholinergic burden of antiparkinsonian therapy, and may worsen the cognitive and autonomic burdens of the illness. Therefore, randomized controlled trials (RCTs) are needed to optimize treatment paradigms for urinary symptoms in PD.

The investigators propose a three-site, RCT conducted at the Atlanta (lead site), Birmingham and Richmond VA's to establish non-inferiority of pelvic floor muscle exercise-based behavioral therapy compared to drug therapy for OAB symptoms in adults with PD. Groups will be stratified by OAB symptom severity, PD motor symptom severity, gender, and site. The investigators will randomize 90 participants in order to complete the study in 80 participants, assuming 85% power and a non-inferiority margin for the OAB symptom score of 15% at 12-weeks. The primary outcome measure will be urinary symptom severity as measured by the International Consultation on Incontinence Questionnaire (ICIQ)-OAB symptom score collected at 3 time points during the study: baseline, 6 weeks, and 12 weeks. The investigators' benchmark for successful treatment will be a 2 point reduction in the ICIQ-OAB symptom score, which corresponds with perceived benefit in preliminary studies of behavioral therapy treatment for OAB symptoms in PD. To evaluate the primary efficacy outcome, the investigators will utilize a random effects mixed model and adjust for baseline OAB symptom score severity. Additionally, in order to better understand central control mechanisms of bladder function, the investigators will determine if domain-specific cognitive function impacts the response to exercise-based behavioral therapy or drug therapy for urinary symptoms. At baseline and 12 weeks, randomized participants will undergo a brief neuropsychological battery. Understanding how domain-specific cognitive function impacts response to treatment may inform new targets for rehabilitation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PD determined by a board-certified neurologist with specialty training in movement disorders
* An ICIQ-OAB Symptom Score of 7, which indicates clinically significant symptoms of OAB, defined as presence of urinary urgency with or without urgency incontinence usually with increased daytime frequency and nocturia in the absence of infection or other obvious pathology

Exclusion Criteria:

* Significant cognitive impairment, as indicated by a Montreal Cognitive Assessment (MoCA) score of < 18, which is the recommended diagnostic cutpoint for dementia in PD.
* Previous intensive pelvic floor muscle exercise training
* Clinically significant depression as measured by a Geriatric Depression Scale-Short Form score 10 which could affect motivation to fully engage in the intervention
* Use of an indwelling urinary catheter
* Post-void residual (PVR) urine measurement by bladder ultrasound of 150 mL
* Severe uterine prolapse past the vaginal introitus
* Poorly controlled diabetes defined by a hemoglobin A1c (HgbA1c) of >9.0% within the last 3 months. Participants with poorly controlled diabetes will be offered enrollment if the OAB symptoms persist after improvement in diabetes control
* Chronic renal failure and on hemodialysis
* Genitourinary cancer with ongoing surgical or external beam radiation treatment
* Previous artificial urinary sphincter, sling procedure or implanted sacral neuromodulation device
* History of bladder-injection of botulinum toxin in the last 12 months
* Any unstable health condition expected to result in hospitalization or death within in the next 3 months as determined by site principal investigator.
* Hypersensitivity to drug class
* Contraindication to the study drug (solifenacin) including: narrow angle glaucoma, history of gastric retention, history of acute urinary retention requiring catheterization
* Current use of a bladder relaxant - permitted to enroll after two week washout
* Hematuria on microscopic examination in the absence of infection. A urologic consultation will be recommended and enrollment will depend on clearance by a urologist and agreement by the site PI that entry into the treatment protocol is not contraindicated
* If on diuretic, dose should be stable for at least 4 weeks
* If taking an alpha-blocker, dose should be stable for at least 4 weeks
* If taking dutasteride or finasteride, dose should be stable for at least 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Camille Vaughan, MD MS, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (4):
- United States (4):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying publications resulting from the proposed research will be shared outside VA through a de-identified, anonymized Dataset under a written agreement that adheres to any applicable Informed Consent provisions and prohibits the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.

REFERENCES:
- [Derived] Vaughan CP, Morley JF, Lehosit J, McGwin G, Muirhead L, Khakharia A, Johnson TM 2nd, Evatt ML, Sergent T, Burgio KL, Markland AD. Behavioral Compared With Drug Therapy for Overactive Bladder Symptoms in Parkinson Disease: A Randomized Noninferiority Trial. JAMA Neurol. 2025 Sep 1;82(9):925-931. doi: 10.1001/jamaneurol.2025.1904. PMID 40658410

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Therapy | Drug Therapy
Started | 36 | 41
Completed | 36 | 37
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Therapy | Drug Therapy | Total
Number analyzed (Participants) | 36 | 41 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (9.3) | 72.9 (8.4) | 71.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 29 | 36 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 37 | 69
  Black | 2 | 1 | 3
  Other | 2 | 3 | 5
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — Validated measure of cognitive function, 0-30 point scale with higher score indicating better cognitive function
  units on a scale | 24.8 (3.3) | 23.9 (3.1) | 24.3 (3.2)
ICIQ-OAB Symptom Score [Mean (Standard Deviation); unit: units on a scale] — International Consultation on Incontinence Questionnaire - Overactive Bladder Symptom Score, score range 0-16 with higher scores indicating more frequent (worse) urinary symptoms
  units on a scale | 8.5 (1.4) | 9.1 (1.7) | 8.8 (1.5)
ICIQ-OAB QoL [Mean (Standard Deviation); unit: units on a scale] — International Consultation on Incontinence Overactive Bladder Quality of Life scale, range 25-160 with higher scores indicating worse quality of life related to overactive bladder
  units on a scale | 72.5 (22.8) | 69.8 (27.3) | 71.2 (25.0)
Bladder-diary derived daily incontinence [Mean (Standard Deviation); unit: incontinence episodes per day] | 1.29 (1.90) | 0.97 (1.71) | 1.12 (1.80)

OUTCOME MEASURES:

1. Primary Outcome: ICIQ-OAB Questionnaire
Description: The ICIQ-OAB questionnaire is a 4-question assessment of OAB symptoms and the degree to which they bother the respondent (urgency, frequency, nocturia, UI).
Time Frame: ICIQ-OAB Symptom score at 12 weeks
Population: Multiple imputation methods used to account for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Therapy | Drug Therapy
Number analyzed (Participants) | 36 | 41
score on a scale | 5.5 (2.0) | 5.8 (2.4)

2. Secondary Outcome: Bladder Diary
Description: 7-day bladder diary includes daily participant-reported incontinence episodes
Time Frame: Incontinence episodes per day at 12 weeks
Measure: Mean (Standard Deviation); unit: Incontinence episodes per day
Arm/Group | Behavioral Therapy | Drug Therapy
Number analyzed (Participants) | 21 | 27
Incontinence episodes per day | 0.45 (1.19) | 0.86 (1.48)

3. Secondary Outcome: ICIQ-OAB QOL
Description: Assessment of quality of life related to the impact of overactive bladder symptoms on daily activities, range 25-160 with higher scores indicating worse quality of life related to overactive bladder
Time Frame: ICIQ-OAB QOL score at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Therapy | Drug Therapy
Number analyzed (Participants) | 36 | 41
units on a scale | 56.6 (22.2) | 56.8 (26.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Behavioral Therapy | Drug Therapy
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/36 | 6/41
Other Adverse Events (participants affected / at risk) | 0/36 | 4/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Therapy (N=36) | Drug Therapy (N=41)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Edema (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Foot sore (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Therapy (N=36) | Drug Therapy (N=41)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT03149809/Prot_SAP_000.pdf